CLINICAL TRIAL: NCT06183060
Title: Department of Anesthesiology, Peking University Third Hospital, Associate Chief Physician; M.D.
Brief Title: Study on the Decision Support System of Difficult Airway Evaluation
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2022105
Record Dates: First submitted 2023-11-20; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-11

CONDITIONS: Difficult Airway
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- difficult laryngoscopy group: Cormack-Lehane (C-L) scale: class III-IV
  Interventions: Procedure: endotracheal intubation
- easy laryngoscopy group: Cormack-Lehane (C-L) scale: class I-II
  Interventions: Procedure: endotracheal intubation

INTERVENTIONS:
Procedure: endotracheal intubation — all patients will receive laryngoscopy and endotracheal intubation

SUMMARY:
Based on the evaluation of preoperative physical indicators and radiologic indicators of cervical surgery, this study puts forward effective indicators for predicting difficult airway before operation, and establishes a comprehensive decision support system of difficult airway evaluation, so as to provide a theoretical basis for the early warning of difficult airway before cervical spondylosis surgery.

DETAILED DESCRIPTION:
In the past, the evaluation of difficult airway mainly depended on physical indicators, but the internal structure of airway could not be found by appearance inspection. Therefore, unexpected emergency airway often appeared in clinical work, which seriously affected medical safety. In this study, the specific mechanism of difficult laryngoscopy in patients undergoing cervical spondylosis surgery is clarified by the combination of the physical indicators and radiologic indicators. On this basis, we will establish the preoperative airway evaluation system for cervical spondylosis surgery, optimize the standardized process of preoperative airway evaluation, and accurately screen out high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* patients of ASA I-III
* scheduled for elective surgery for cervical spondylosis under general anesthesia with tracheal intubation

Exclusion Criteria:

* patients with cervical spine instability
* oropharyngeal mass
* airway disease
* preoperative imaging data were incomplete
* refuse to sign informed consent

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective cervical spine surgery for cervical spondylosis (spinal cord and nerve root type
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Cormack-Lehane (CL) classification | During induction
  describe laryngeal view during direct laryngoscopy

SECONDARY OUTCOMES:
X1(X-ray indicators) | During review the X-ray image
  distance between the temporomandibular joint and tip of the upper incisors
X2(X-ray indicators) | During review the X-ray image
  perpendicular distance from the hard palate to the tip of the upper incisors
X3(X-ray indicators) | During review the X-ray image
  length of the mandibular body
X4(X-ray indicators) | During review the X-ray image
  vertical distance from the highest point of the hyoid bone to the mandibular body
X5(X-ray indicators) | During review the X-ray image
  distance from the antero-inferior border of the fourth cervical vertebra to the antero-superior border of the ﬁrst cervical vertebra
X6(X-ray indicators) | During review the X-ray image
  atlanto-occipital gapantero-superior border of the ﬁrst cervical vertebra
X7(X-ray indicators) | During review the X-ray image
  horizontal distance from the highest point of the hyoid bone to the border of the nearest cervical vertebra
X8(X-ray indicators) | During review the X-ray image
  distance between the spinous processes of the ﬁrst cervical vertebra and the second cervical vertebra
A1 (X-ray indicators) | During review the X-ray image
  the angle between a line passing through the bottom of second cervical vertebra and a line passing through the bottom of sixth cervical vertebra in the neutral/ extension position
Hp-h (CT/MRI indicators) | During review the CT/MRI image
  the distance from back end of the hard palate to the top of hyoid
Ht (CT/MRI indicators) | During review the CT/MRI image
  the height of the tongue base, along Hp-h from the tongue to the top of hyoid
Dt-p (CT/MRI indicators) | During review the CT/MRI image
  the distance from the back end of tongue to posterior pharyngeal wall
Dt (CT/MRI indicators) | During review the CT/MRI image
  the distance from the back end of tongue to Hp-h
S (CT/MRI indicators) | During review the CT/MRI image
  the central sectional area of the tongue base behind Hp-h
W (CT/MRI indicators) | During review the CT/MRI image
  the maximal width of the tongue base
V (CT/MRI indicators) | During review the CT/MRI image
  volume of the tongue base
Rs (CT/MRI indicators) | During review the CT/MRI image
  Rs= S/( Hp-h* Dt-p); Rv =V/( Hp-h* Dt-p*W)
MRI1 (MRI indicators) | During review the CT/MRI image
  distance between the base of the tongue and the posterior pharyngeal wall
MRI2 (MRI indicators) | During review the CT/MRI image
  distance between the epiglottis and the posterior pharyngeal wall
MRI3 (MRI indicators) | During review the CT/MRI image
  distance between the uvula and the posterior pharyngeal wall
MRI4 (MRI indicators) | During review the CT/MRI image
  distance between the vocal cords and the posterior pharyngeal wall
MRI5 (MRI indicators) | During review the CT/MRI image
  length of the epiglottis

OTHER OUTCOMES:
inter-incisor gap | measurement one day before operation]
  physical indicator
thyromental distance | measurement one day before operation]
  physical indicator
neck circumference, | measurement one day before operation]
  physical indicator
modified Mallampati test, | measurement one day before operation]
  physical indicator

CONTACTS AND LOCATIONS:
Overall Officials: Yongzheng Han, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
if necessary, access the data by contacting the project leader
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after the project finished and manuscript published
Access Criteria: contact the project leader and data can only be used for scientific research

REFERENCES:
- [Result] Han YZ, Tian Y, Xu M, Ni C, Li M, Wang J, Guo XY. Neck circumference to inter-incisor gap ratio: a new predictor of difficult laryngoscopy in cervical spondylosis patients. BMC Anesthesiol. 2017 Apr 4;17(1):55. doi: 10.1186/s12871-017-0346-y. PMID 28376741
- [Result] Han YZ, Tian Y, Zhang H, Zhao YQ, Xu M, Guo XY. Radiologic indicators for prediction of difficult laryngoscopy in patients with cervical spondylosis. Acta Anaesthesiol Scand. 2018 Apr;62(4):474-482. doi: 10.1111/aas.13078. Epub 2018 Jan 31. PMID 29388207